CLINICAL TRIAL: NCT02975349
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Study of M2951 With a Parallel, Open-Label, Active Control Group (Tecfidera), in Patients With Relapsing Multiple Sclerosis to Evaluate Efficacy, Safety, Tolerability, Pharmacokinetics, and Biological Activity.
Brief Title: A Study of Efficacy and Safety of M2951 in Participants With Relapsing Multiple Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Results from the EVOLUTION clinical trials showed evobrutinib did not meet its primary endpoint of annualized relapse rate for up to 156 weeks compared to oral teriflunomide in both studies.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS200527-0086; 2016-001448-21 (EudraCT Number)
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: M2951; Relapsing Multiple Sclerosis; Bruton's Tyrosine Kinase inhibitor
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — evobrutinib; Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo then Evobrutinib 25 mg QD (Period 2) (Experimental): Participants who received placebo matched to Evobrutinib tablet orally for 24 weeks in active treatment period 1 received Evobrutinib 25 milligram (mg) orally, once daily (QD) in blinded extension (BE) period from week 25 to week 48.
  Interventions: Drug: Evobrutinib
- Evobrutinib 25 mg QD (Period 1, 2 and 3) (Experimental): Participants received Evobrutinib 25 mg orally, QD up to Week 48 in active treatment period 1 and BE period received Evobrutinib 25 mg QD orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
  Interventions: Drug: Evobrutinib
- Evobrutinib 75 mg QD (Period 1, 2 and 3) (Experimental): Participants received Evobrutinib 75 mg orally, QD up to Week 48 in active treatment period 1 and BE period received Evobrutinib 75 mg QD orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
  Interventions: Drug: Evobrutinib
- Evobrutinib 75 mg BID (Period 1, 2 and 3) (Experimental): Participants received Evobrutinib 75 mg orally, twice daily (BID) up to Week 48 in active treatment period 1 and BE period received Evobrutinib 75 mg BID orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
  Interventions: Drug: Evobrutinib
- Tecfidera (Period 1, 2 and 3) (Active Comparator): Participants received Tecfidera 120 mg twice daily (BID) for first 7 days followed by 240 mg orally, BID up to Week 48 in active treatment period 1 and BE period received Tecfidera 120 mg BID orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
  Interventions: Drug: Tecfidera
- Placebo (Placebo Comparator): Participants received placebo matched to Evobrutinib tablet orally for 24 weeks in active treatment period 1.
  Interventions: Drug: Placebo
- Placebo + Evobrutinib 25 mg QD (Period 3) (Experimental): Participants who received placebo matched to Evobrutinib tablet orally for 24 weeks in active treatment period 1 received Evobrutinib 25 mg orally, QD from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
  Interventions: Drug: Evobrutinib

INTERVENTIONS:
Drug: Evobrutinib — Participants received Evobrutinib 75 mg orally, QD up to Week 48 in active treatment period 1 and BE period received Evobrutinib 75 mg QD orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
  Other Names: M2951
  Arms: Evobrutinib 75 mg BID (Period 1, 2 and 3)
Drug: Evobrutinib — Participants received Evobrutinib 25 mg orally, QD up to Week 48 in active treatment period 1 and BE period received Evobrutinib 25 mg QD orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
  Other Names: M2951
  Arms: Evobrutinib 25 mg QD (Period 1, 2 and 3); Placebo + Evobrutinib 25 mg QD (Period 3); Placebo then Evobrutinib 25 mg QD (Period 2)
Drug: Evobrutinib — Participants received Evobrutinib 75 mg orally, QD up to Week 48 in active treatment period 1 and BE period received Evobrutinib 75 mg QD orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
  Other Names: M2951
  Arms: Evobrutinib 75 mg QD (Period 1, 2 and 3)
Drug: Placebo — Placebo were administered for 24 weeks in active treatment period.
  Arms: Placebo
Drug: Tecfidera — Participants received Tecfidera 120 mg twice daily (BID) for first 7 days followed by 240 mg orally, BID up to Week 48 in active treatment period 1 and BE period received Tecfidera 120 mg BID orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
  Arms: Tecfidera (Period 1, 2 and 3)

SUMMARY:
The aim of this protocol is to find out about the safety and effectiveness of M2951 in participants with relapsing multiple sclerosis. Participants were placed into 1 of 3 groups to receive M2951, placebo or tecfidera for 24 weeks. After 24 weeks, the participants on placebo were given M2951.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of relapsing multiple sclerosis (may include participants with Secondary Progressive Multiple Sclerosis (SPMS) with superimposed relapses provided they meet the other criteria) in accordance with revised McDonald criteria for MS and Lublin and Reingold
* Male or female aged 18 to 65 years
* One or more documented relapses within the 2 years before Screening with either: a) One relapse which occurred within the last year prior to randomization or b) the presence of at least 1 gadolinium-positive (Gd+) T1 lesion within 6 months prior to randomization would make the patient eligible.
* Expanded Disability Status Scale score of 0 to 6 at Baseline
* Women of childbearing potential must use a supplementary barrier method together with a highly effective method of contraception (according to International Council for Harmonisation [ICH] guidance M3[R2]) for 4 weeks prior to randomization, throughout the trial, and for 90 days after the last dose of IMP.
* Signed and dated informed consent (participant must be able to understand the informed consent) indicating that the participant has been informed of all the pertinent aspects of the trial prior to enrolment and will comply with the requirements of the protocol.

Exclusion Criteria:

* Progressive MS
* Disease duration > 15 years in participants with EDSS of 2 or less
* Use of the following, as determined in the protocol ; rituximab, ocrelizumab, mitoxantrone, or lymphocyte-depleting therapies, lymphocyte trafficking blockers (eg, natalizumab, fingolimod), intravenous (IV) immunoglobulins (Ig), plasmapheresis, immunosuppressive treatments, B-interferons or glatiramer acetate, Systemic glucocorticoids, teriflunomide
* Exposure to Tecfidera within 6 months prior to randomization
* Any allergy, contraindication, or inability to tolerate Tecfidera
* Treatment with dalfampridine (fampridine, Ampyra) unless on a stable dose for ≥ 30 days prior to randomization
* Inability to comply with MRI scanning
* Immunologic disorder other than MS, with the exception of secondary well-controlled diabetes or thyroid disorder, or any other condition requiring oral, IV, intramuscular, or intra-articular corticosteroid therapy
* Vaccination with live or live-attenuated virus vaccine within 1 month prior to Screening
* Severe drug allergy or history of anaphylaxis, or allergy to the IMP or any of its incipients
* Active, clinically significant viral, bacterial, or fungal infection, or any major episode of infection requiring hospitalization or treatment with parenteral anti-infectives within 4 weeks of Screening, or completion of oral anti-infectives within 2 weeks before or during Screening, or a history of recurrent infections (ie, 3 or more of the same type of infection in a 12-month rolling period). Vaginal candidiasis, onychomycosis, and genital or oral herpes simplex virus considered by the Investigator to be sufficiently controlled would not be exclusionary.
* History of or positive testing for human immunodeficiency virus (HIV), hepatitis C (HCV) antibody and/or polymerase chain reaction, hepatitis B surface antigen (HBsAg) (+) and/or hepatitis B core total, and/or immunoglobulin M (IgM) antibody (+) at Screening.
* The participant: • Has a history of or current diagnosis of active tuberculosis (TB) or • Is currently undergoing treatment for latent TB infection (LTBI) or • Has an untreated LTBI or • Has a positive QuantiFERON®-TB test at Screening.
* Indeterminate QuantiFERON®
* Participants with current household contacts with active TB will also be excluded
* History of splenectomy or any major surgery within 2 months prior to Screening
* History of myocardial infarction or cerebrovascular event as per the protocol
* History of attempted suicide within 6 months prior to Screening or a positive response to items 4 or 5 of Columbia-Suicide Severity Rating Scale (C-SSRS)
* An episode of major depression within the last 6 months prior to Screening
* On anticoagulation, fish oil supplements, or antiplatelet therapy other than daily aspirin for cardioprotection and treatment of Tecfidera induced flushing
* History of cancer, except adequately treated basal cell or squamous cell carcinoma of the skin
* Breastfeeding/lactating or pregnant women
* Participation in any investigational drug trial within 1 month or 5 half-lives of the investigational drug, whichever is longest, prior to Screening
* Participants currently receiving (or unable to stop using prior to receiving the first dose of IMP) medications or herbal supplements known to be potent inhibitors of cytochrome P450 3A (CYP3A)
* History of or current alcohol or substance abuse
* Clinically significant abnormality on electrocardiogram or screening chest X-ray
* Clinically significant laboratory abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (42):
- Bulgaria (6):
  - Research Site, Blagoevgrad
  - Research Site, Dupnitsa
  - Research Site 1, Pleven
  - Research Site 2, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Prague
  - Research Site, Teplice
- Poland (9):
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Oświęcim
  - Research Site, Plewiska
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Warsaw
- Russia (6):
  - Research Site, Kazan'
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Saransk
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Užice
- Slovakia (3):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Dubnica nad Váhom
- Spain (2):
  - Research Site, A Coruña
  - Research Site, Barcelona
- Ukraine (7):
  - Research Site, Chernivtsi
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Poltava
  - Research Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
Per company policy and with respect to the principles set forth by the International Federation of Pharmaceutical Manufacturers and Associations (IFPMA), the European Federation of Pharmaceutical Industries and Associations (EFPIA), the Pharmaceutical Research and Manufacturers of America (PhRMA), the Declaration of Helsinki, and applicable laws and regulations , we inform the public about the designs and results of our clinical trials in a timely and balanced manner, regardless of the outcome. We are committed to enhancing public health through responsible sharing of clinical trial data in a manner that is consistent with: safeguarding the privacy of patients; respecting the integrity of national regulatory systems; and maintaining incentives for investment in biomedical research.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the occurrence of an approval of a new product or a new indication for an approved product in both the European Union and the United States after January 1, 2014 If approval of a product is not sought, Merck shall make publicly available such data within eighteen months after the trial completion date. Data will not be shared for products and indications approved prior to January 1, 2014
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researcher qualifications and legitimacy of the research purpose.
URL: https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- [Result] Montalban X, Arnold DL, Weber MS, Staikov I, Piasecka-Stryczynska K, Willmer J, Martin EC, Dangond F, Syed S, Wolinsky JS; Evobrutinib Phase 2 Study Group. Placebo-Controlled Trial of an Oral BTK Inhibitor in Multiple Sclerosis. N Engl J Med. 2019 Jun 20;380(25):2406-2417. doi: 10.1056/NEJMoa1901981. Epub 2019 May 10. PMID 31075187
- [Result] Arnold DL, Elliott C, Martin EC, Hyvert Y, Tomic D, Montalban X. Effect of Evobrutinib on Slowly Expanding Lesion Volume in Relapsing Multiple Sclerosis: A Post Hoc Analysis of a Phase 2 Trial. Neurology. 2024 Mar 12;102(5):e208058. doi: 10.1212/WNL.0000000000208058. Epub 2024 Feb 9. PMID 38335474
- [Result] Papasouliotis O, Mitchell D, Girard P, Dangond F, Dyroff M. Determination of a clinically effective evobrutinib dose: Exposure-response analyses of a phase II relapsing multiple sclerosis study. Clin Transl Sci. 2022 Dec;15(12):2888-2898. doi: 10.1111/cts.13407. Epub 2022 Sep 30. PMID 36126241
- [Result] Montalban X, Wallace D, Genovese MC, Tomic D, Parsons-Rich D, Le Bolay C, Kao AH, Guehring H. Characterisation of the safety profile of evobrutinib in over 1000 patients from phase II clinical trials in multiple sclerosis, rheumatoid arthritis and systemic lupus erythematosus: an integrated safety analysis. J Neurol Neurosurg Psychiatry. 2023 Jan;94(1):1-9. doi: 10.1136/jnnp-2022-328799. Epub 2022 Nov 23. PMID 36418156
- [Result] Bar-Or A, Cross AH, Cunningham AL, Hyvert Y, Seitzinger A, Guhring H, Drouin EE, Alexandri N, Tomic D, Montalban X. Antibody response to SARS-CoV-2 vaccines in patients with relapsing multiple sclerosis treated with evobrutinib: A Bruton's tyrosine kinase inhibitor. Mult Scler. 2023 Oct;29(11-12):1471-1481. doi: 10.1177/13524585231192460. Epub 2023 Aug 25. PMID 37626477
- [Derived] Montalban X, Wallace D, Genovese MC, Tomic D, Parsons-Rich D, Bolay CL, Kao AH, Guehring H. A plain language summary of what clinical studies can tell us about the safety of evobrutinib - a potential treatment for multiple sclerosis. Neurodegener Dis Manag. 2023 Aug;13(4):207-213. doi: 10.2217/nmt-2023-0003. Epub 2023 Jun 22. PMID 37345645
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527-0086
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Period 1): Participants received placebo matched to Evobrutinib tablet orally for 24 weeks in active treatment period 1.
Period: Active Treatment Period (24 Weeks)
Arm/Group | Placebo (Period 1) | Placebo Then Evobrutinib 25 mg QD (Period 2) | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Started | 54 | 0 | 0 | 52 | 53 | 54 | 54
Safety Analysis Set (Safety analysis set included all participants who received at least 1 dose of evobrutinib or placebo or Tecfidera.) | 54 | 0 | 0 | 52 | 53 | 54 | 54
Completed | 49 | 0 | 0 | 47 | 48 | 48 | 52
Not Completed | 5 | 0 | 0 | 5 | 5 | 6 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 2 | 2 | 6 | 2
Period: Blinded Extension Period (24 Weeks)
Arm/Group | Placebo (Period 1) | Placebo Then Evobrutinib 25 mg QD (Period 2) | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Started | 0 | 49 | 0 | 47 | 48 | 48 | 52
Completed | 0 | 42 | 0 | 43 | 44 | 46 | 52
Not Completed | 0 | 7 | 0 | 4 | 4 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 0 | 2 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Open-label Extension Period (336 Weeks)
Arm/Group | Placebo (Period 1) | Placebo Then Evobrutinib 25 mg QD (Period 2) | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Started | 0 | 0 | 39 | 39 | 42 | 44 | 49
Completed | 0 | 0 | 28 | 25 | 33 | 35 | 39
Not Completed | 0 | 0 | 11 | 14 | 9 | 9 | 10
Not completed — Adverse Event | 0 | 0 | 3 | 2 | 2 | 1 | 2
Not completed — Study reached its predefined end | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — COVID-19 Related | 0 | 0 | 0 | 1 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 3 | 3 | 1 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 7 | 2 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Modified Intent-To-Treat (mITT) analysis set included participants who belong to both Intent To Treat (ITT, consisted all participants who randomly allocated to a treatment, based on the intention to treat "as randomized" principle) and safety analysis sets (consisted all participants who receive at least 1 dose of trial treatment), and who have at least one baseline and one post-baseline magnetic resonance imaging (MRI) assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3) | Total
Number analyzed (Participants) | 53 | 50 | 51 | 53 | 54 | 261
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (10.77) | 42.4 (9.37) | 42.9 (10.07) | 42.2 (11.50) | 42.8 (11.70) | 42.4 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 32 | 35 | 36 | 39 | 181
  Male | 14 | 18 | 16 | 17 | 15 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 2 | 5
  Not Hispanic or Latino | 52 | 49 | 51 | 52 | 52 | 256
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 53 | 50 | 51 | 53 | 54 | 261
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Gadolinium-Enhancing T1 Lesions
Description: Analysis of T1-Gadolinium enhancing lesions was done using magnetic resonance imaging (MRI) scans. As per planned analysis, Tecfidera treatment group was not included in inferential analysis.
Time Frame: Week 12 to Week 24
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 53 | 50 | 51 | 53 | 54
Lesions | 3.85 (5.436) | 4.06 (8.024) | 1.69 (4.693) | 1.15 (3.702) | 4.78 (22.045)
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Evobrutinib 25 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.2947, Negative Binomial model; Lesion rate ratio = 1.45, 95% CI 2-sided [0.72 to 2.91]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.0015, Negative Binomial model; Lesion rate ratio = 0.30, 95% CI 2-sided [0.14 to 0.63]
Statistical Analysis 3: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg BID (Period 1, 2 and 3); Test type: Superiority; p = 0.0313, Negative Binomial model; Lesion rate ratio = 0.44, 95% CI 2-sided [0.21 to 0.93]

2. Secondary Outcome: Annualized Relapse Rate (ARR) at Week 24
Description: A qualifying relapse is defined as new, worsening or recurrent neurological symptoms attributed to Multiple Sclerosis (MS) that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. As per planned analysis, Tecfidera treatment group was not included in inferential analysis.
Time Frame: Week 24
Population: The modified ITT (mITT) analysis set consists of all participants who belong to both the ITT and safety analysis sets, and who have at least one baseline and one post-baseline magnetic resonance imaging (MRI) assessment.
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 53 | 50 | 51 | 53 | 54
relapses per year | 0.37 [0.17 to 0.70] | 0.57 [0.30 to 0.97] | 0.13 [0.03 to 0.38] | 0.08 [0.01 to 0.30] | 0.20 [0.06 to 0.47]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Evobrutinib 25 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.2692, Negative Binomial model; Qualified relapse rate ratio = 1.66, 95% CI 2-sided [0.67 to 4.09]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.0896, Negative Binomial model; Qualified relapse rate ratio = 0.31, 95% CI 2-sided [0.08 to 1.20]
Statistical Analysis 3: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg BID (Period 1, 2 and 3); Test type: Superiority; p = 0.0633, Negative Binomial model; Qualified relapse rate ratio = 0.23, 95% CI 2-sided [0.05 to 1.09]

3. Secondary Outcome: Qualified Relapse-Free Status at Week 24
Description: A qualifying relapse is defined as new, worsening or recurrent neurological symptoms attributed to Multiple Sclerosis (MS) that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. Percentage of participants with qualified relapse-free status at week 24 were reported. As per planned analysis, Tecfidera treatment group was not included in inferential analysis.
Time Frame: Week 24
Population: mITT analysis set consists of all participants who belong to both the ITT and safety analysis sets, and who have at least one baseline and one post-baseline MRI assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 53 | 50 | 51 | 53 | 54
percentage of participants | 77.4 [63.8 to 87.7] | 74.0 [59.7 to 85.4] | 88.2 [76.1 to 95.6] | 86.8 [74.7 to 94.5] | 88.9 [77.4 to 95.8]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Evobrutinib 25 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.5609, Logistic model; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.29 to 1.95]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.0689, Logistic model; Odds Ratio (OR) = 2.79, 95% CI 2-sided [0.92 to 8.41]
Statistical Analysis 3: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg BID (Period 1, 2 and 3); Test type: Superiority; p = 0.1767, Logistic model; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.72 to 5.99]

4. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) at Week 24
Description: The EDSS is an ordinal clinical rating scale in half-point increments. It assesses the following eight functional systems, areas of the central nervous system that control bodily functions: Pyramidal (ability to walk), Cerebellar (coordination), Brain stem (speech and swallowing), Sensory (touch and pain), Bowel and bladder functions, Visual, Mental, Other (includes any other neurological findings due to Multiple Sclerosis [MS]). EDSS overall score ranging from 0 (normal) to 10 (death due to MS). As per planned analysis, Tecfidera treatment group was not included in inferential analysis.
Time Frame: Baseline, Week 24
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 53 | 50 | 51 | 53 | 54
Units on a scale | -0.03 (0.301) | 0.02 (0.622) | -0.14 (0.664) | 0.04 (0.216) | 0.02 (0.274)
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Evobrutinib 25 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.4070, Wilcoxon rank-sum test; Hodges-Lehmann estimate = 0.00, 95% CI 2-sided [0.00 to 0.00]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.5829, Wilcoxon rank-sum test; Hodges-Lehmann estimate = 0.00, 95% CI 2-sided [0.00 to 0.00]
Statistical Analysis 3: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg BID (Period 1, 2 and 3); Test type: Superiority; p = 0.2732, Wilcoxon rank-sum test; Hodges-Lehmann estimate = 0.00, 95% CI 2-sided [0.00 to 0.00]

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs Leading to Death
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the study drug. An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent adverse events are defined as any adverse event with a start date on or after the date of first dose and within 28 days after the date of last dose in the study. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Safety Follow-up (Week 52)
Population: The safety analysis set included of all participants who received at least 1 dose of evobrutinib or placebo or Tecfidera.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 1) | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 54 | 49 | 52 | 53 | 54 | 54
Participants
  TEAEs | 24 | 19 | 28 | 35 | 34 | 35
  Serious TEAEs | 2 | 0 | 2 | 2 | 4 | 2
  TEAEs Leading to Death | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs and Electrocardiograms (ECGs)
Description: Vital signs, including semi supine blood pressure, pulse rate, respiratory rate, weight, and oral temperature were assessed. ECG parameters included rhythm, ventricular rate, PR interval, QRS duration, and QT interval. Number of participants with clinically significant change from baseline in vital signs and ECG were reported. Clinical Significance was decided by the investigator.
Time Frame: Baseline up to Safety Follow-up (Week 52)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 1) | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 54 | 49 | 52 | 53 | 54 | 54
Participants
  Vital Sign Abnormalities | 0 | 0 | 0 | 0 | 0 | 0
  ECG Abnormalities | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Grade 3 or Higher Hematology, Biochemistry and Urinalysis Values
Description: Hematology, biochemistry, and urinalysis values were graded with National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 toxicity grades (where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening and Grade 5 = death). For the hematology and biochemistry parameters, participants with a value grade 3 or higher were reported. For the urinalysis parameters, participants with a value grade 3 or higher, or a value >= 2 upper limit of normal (ULN), or a value classified as ++ Increasing were reported.
Time Frame: Baseline up to Safety Follow-up (Week 52)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 1) | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 54 | 49 | 52 | 53 | 54 | 54
Participants
  Grade >= 3 hematology values | 0 | 2 | 0 | 1 | 0 | 1
  Grade >= 3 biochemistry values | 2 | 8 | 6 | 9 | 16 | 9
  Grade >= 3 or value >= 2 ULN or ++ Increasing urinalysis values | 0 | 2 | 1 | 2 | 2 | 6

8. Secondary Outcome: Absolute Concentrations of Immunoglobulin (Ig) Levels (Active Treatment Period)
Description: Absolute Concentrations serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline (Day 1), Weeks 4, 16, and 24
Population: The safety analysis set included of all participants who received at least 1 dose evobrutinib or placebo or Tecfidera. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Mean (Standard Deviation); unit: Gram per Liter
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 54 | 52 | 53 | 54 | 54
Gram per Liter
  Ig A, Day 1: number analyzed (Participants) | 54 | 51 | 53 | 54 | 54
  Ig A, Day 1 | 1.99 (0.777) | 1.89 (0.764) | 1.90 (0.722) | 1.87 (0.675) | 2.03 (0.763)
  Ig A, Week 4 | 1.98 (0.777) | 1.92 (0.770) | 1.93 (0.762) | 1.94 (0.748) | 1.90 (0.699)
  Ig A, Week 16: number analyzed (Participants) | 53 | 50 | 49 | 53 | 52
  Ig A, Week 16 | 2.07 (0.824) | 2.10 (0.813) | 2.13 (0.832) | 2.08 (0.753) | 2.03 (0.752)
  Ig A, Week 24: number analyzed (Participants) | 50 | 47 | 49 | 48 | 52
  Ig A, Week 24 | 1.99 (0.807) | 2.12 (0.833) | 2.09 (0.838) | 2.09 (0.793) | 1.97 (0.757)
  Ig G, Day 1: number analyzed (Participants) | 54 | 51 | 53 | 54 | 54
  Ig G, Day 1 | 9.61 (1.897) | 9.43 (2.126) | 9.81 (1.841) | 9.62 (1.960) | 9.47 (1.839)
  Ig G, Week 4 | 9.64 (2.094) | 9.34 (1.972) | 9.79 (1.910) | 9.64 (1.987) | 9.05 (1.922)
  Ig G, Week 16: number analyzed (Participants) | 53 | 50 | 49 | 53 | 52
  Ig G, Week 16 | 9.68 (2.085) | 9.41 (2.077) | 9.70 (1.991) | 9.56 (2.129) | 9.58 (1.850)
  Ig G, Week 24: number analyzed (Participants) | 50 | 47 | 49 | 48 | 52
  Ig G, Week 24 | 9.66 (2.081) | 9.46 (2.123) | 9.62 (2.048) | 9.36 (1.988) | 9.27 (1.866)
  Ig M, Day 1: number analyzed (Participants) | 54 | 51 | 53 | 54 | 54
  Ig M, Day 1 | 1.42 (0.692) | 1.27 (0.542) | 1.44 (0.716) | 1.33 (0.684) | 1.27 (0.589)
  Ig M, Week 4: number analyzed (Participants) | 54 | 51 | 53 | 54 | 54
  Ig M, Week 4 | 1.40 (0.668) | 1.21 (0.526) | 1.32 (0.654) | 1.28 (0.656) | 1.23 (0.603)
  Ig M, Week 16: number analyzed (Participants) | 53 | 50 | 49 | 53 | 52
  Ig M, Week 16 | 1.43 (0.703) | 1.13 (0.558) | 1.24 (0.639) | 1.20 (0.689) | 1.28 (0.678)
  Ig M, Week 24: number analyzed (Participants) | 49 | 47 | 49 | 48 | 52
  Ig M, Week 24 | 1.44 (0.748) | 1.03 (0.499) | 1.20 (0.672) | 1.08 (0.494) | 1.29 (0.667)

9. Secondary Outcome: Absolute Concentrations of Immunoglobulin (Ig) Levels (Blinded Extension Period)
Description: Absolute Concentrations serum levels of IgG, IgA, IgM were assessed.
Time Frame: Week 48
Population: The safety analysis set included of all participants who received at least 1 dose evobrutinib or placebo or Tecfidera. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure. Results reported are for blinded extension period only and no participants took placebo during this period.
Measure: Mean (Standard Deviation); unit: Gram per Liter
Arm/Group | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 50 | 51 | 54 | 52
Gram per Liter
  IgA | 2.13 (0.807) | 2.18 (0.790) | 2.23 (0.838) | 2.06 (0.695)
  IgG | 9.53 (2.070) | 9.74 (1.902) | 9.38 (2.189) | 9.60 (1.968)
  IgM | 1.08 (0.557) | 1.13 (0.639) | 1.10 (0.692) | 1.28 (0.635)

10. Secondary Outcome: Change From Baseline in Immunoglobulin (Ig) Levels (Active Treatment Period)
Description: Change from baseline in the serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline (Day 1), Weeks 4, 16, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Gram per Liter
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 54 | 50 | 53 | 54 | 54
Gram per Liter
  Ig A, Week 4 | -0.02 (0.201) | 0.02 (0.165) | 0.04 (0.169) | 0.07 (0.195) | -0.13 (0.238)
  Ig A, Week 16: number analyzed (Participants) | 51 | 48 | 49 | 53 | 52
  Ig A, Week 16 | 0.10 (0.188) | 0.18 (0.245) | 0.21 (0.313) | 0.22 (0.209) | -0.02 (0.274)
  Ig A, Week 24: number analyzed (Participants) | 49 | 44 | 48 | 48 | 52
  Ig A, Week 24 | 0.06 (0.250) | 0.21 (0.283) | 0.18 (0.416) | 0.22 (0.229) | -0.06 (0.207)
  Ig G, Week 4 | 0.02 (0.758) | -0.10 (0.697) | -0.02 (0.688) | 0.02 (0.581) | -0.42 (0.926)
  Ig G, Week 16: number analyzed (Participants) | 53 | 48 | 49 | 53 | 52
  Ig G, Week 16 | 0.04 (0.747) | -0.07 (0.964) | -0.10 (1.068) | -0.05 (0.710) | 0.07 (0.961)
  Ig G, Week 24: number analyzed (Participants) | 50 | 45 | 49 | 48 | 52
  Ig G, Week 24 | 0.06 (0.682) | 0.00 (1.228) | -0.15 (1.058) | -0.28 (0.774) | -0.23 (0.882)
  Ig M, Week 4 | -0.01 (0.210) | -0.06 (0.100) | -0.12 (0.233) | -0.05 (0.133) | -0.04 (0.132)
  Ig M, Week 16: number analyzed (Participants) | 53 | 48 | 49 | 53 | 52
  Ig M, Week 16 | 0.02 (0.177) | -0.12 (0.184) | -0.18 (0.244) | -0.14 (0.189) | -0.00 (0.184)
  Ig M, Week 24: number analyzed (Participants) | 50 | 45 | 49 | 48 | 52
  Ig M, Week 24 | 0.04 (0.163) | -0.14 (0.286) | -0.20 (0.289) | -0.21 (0.167) | -0.00 (0.186)

11. Secondary Outcome: Change From Baseline in Immunoglobulin (Ig) Levels (Blinded Extension Period)
Description: Change from baseline in the serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline (Week 25), Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Gram per Liter
Arm/Group | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 48 | 51 | 54 | 52
Gram per Liter
  IgA | 0.26 (0.248) | 0.28 (0.275) | 0.36 (0.320) | 0.03 (0.316)
  IgG | 0.11 (1.024) | -0.08 (0.940) | -0.24 (0.883) | 0.10 (1.244)
  IgM | -0.18 (0.211) | -0.27 (0.287) | -0.23 (0.218) | -0.01 (0.198)

12. Secondary Outcome: Absolute Concentration of B Cells (Active Treatment Period)
Description: Absolute concentration of B Cells are reported.
Time Frame: Baseline (Day 1), Weeks 4, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cells per micro-liter
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 52 | 52 | 53 | 53 | 52
cells per micro-liter
  Day 1: number analyzed (Participants) | 52 | 52 | 49 | 51 | 48
  Day 1 | 242 (134.2) | 208 (117.5) | 247 (131.8) | 219 (113.7) | 210 (97.4)
  Week 4: number analyzed (Participants) | 52 | 50 | 53 | 53 | 52
  Week 4 | 243 (130.8) | 220 (92.7) | 277 (156.2) | 270 (143.2) | 201 (114.3)
  Week 24: number analyzed (Participants) | 49 | 44 | 49 | 47 | 52
  Week 24 | 264 (154.9) | 230 (119.7) | 235 (115.3) | 214 (105.0) | 180 (114.3)

13. Secondary Outcome: Absolute Concentration of B Cells (Blinded Extension Period)
Description: Absolute concentration of B Cells were reported.
Time Frame: Weeks 48 and 52
Population: The safety analysis set included of all participants who received at least 1 dose evobrutinib or placebo or Tecfidera. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signified those participants who were evaluable for the specified category at given time points. Results reported are for blinded extension period only and no participants took placebo during this period.
Measure: Mean (Standard Deviation); unit: cells per micro-liter
Arm/Group | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 49 | 51 | 54 | 47
cells per micro-liter
  Week 48 | 203 (111.9) | 222 (148.8) | 187 (87.1) | 181 (109.8)
  Week 52: number analyzed (Participants) | 6 | 7 | 8 | 2
  Week 52 | 227 (93.7) | 206 (140.3) | 154 (73.6) | 135 (29.0)

14. Secondary Outcome: Change From Baseline in Absolute B Cells (Active Treatment Period)
Description: Change from baseline in absolute B cells are reported.
Time Frame: Baseline (Day 1), Weeks 4 and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cells per micro-liter
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 52 | 50 | 53 | 53 | 52
cells per micro-liter
  Week 4 | -5 (94.5) | 9 (112.2) | 31 (114.2) | 50 (86.7) | -3 (111.0)
  Week 24: number analyzed (Participants) | 49 | 44 | 49 | 47 | 52
  Week 24 | 7 (135.8) | 13 (98.2) | -15 (128.5) | -9 (85.1) | -26 (113.9)

15. Secondary Outcome: Change From Baseline in Absolute B Cells (Blinded Extension Period)
Description: Change from baseline in absolute B cells are reported.
Time Frame: Baseline (Week 25), Weeks 48 and 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: cells per micro-liter
Arm/Group | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 49 | 51 | 54 | 47
cells per micro-liter
  Week 48 | -5 (116.1) | -30 (148.2) | -32 (97.9) | -15 (105.7)
  Week 52: number analyzed (Participants) | 6 | 7 | 8 | 2
  Week 52 | -28 (209.8) | -25 (65.5) | -81 (119.0) | 15 (22.6)

16. Secondary Outcome: Total Number of New Gadolinium-positive (Gd+) T1 Lesions
Description: Analysis of Gadolinium-positive T1 lesions was done using magnetic resonance imaging (MRI) scans. As per planned analysis, Tecfidera treatment group was not included in inferential analysis.
Time Frame: Week 12 to 24
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 53 | 50 | 51 | 53 | 54
Lesions | 3.08 (4.371) | 3.44 (6.846) | 1.20 (3.499) | 0.98 (3.273) | 3.24 (15.320)
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Evobrutinib 25 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.3676, Negative Binomial; Lesion rate ratio = 1.36, 95% CI 2-sided [0.70 to 2.65]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.0005, Negative Binomial; Lesion rate ratio = 0.27, 95% CI 2-sided [0.13 to 0.57]
Statistical Analysis 3: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg BID (Period 1, 2 and 3); Test type: Superiority; p = 0.0157, Negative Binomial; Lesion rate ratio = 0.41, 95% CI 2-sided [0.20 to 0.85]

17. Secondary Outcome: Mean Per-scan Number of Gadolinium-positive (Gd+) T1 Lesions
Description: as for outcome 16
Time Frame: Week 12 to Week 24
Population: mITT analysis set consists of all participants who belong to both the ITT and safety analysis sets, and who have at least one baseline and one post-baseline magnetic resonance imaging (MRI) assessment.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 53 | 50 | 51 | 53 | 54
Lesions | 1.02 (1.439) | 1.31 (3.130) | 0.42 (1.173) | 0.34 (0.960) | 1.45 (7.293)
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Evobrutinib 25 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.9731, Wilcoxon rank-sum test; Hodges-Lehmann estimate = 0.00, 95% CI 2-sided [-0.25 to 0.25]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.0017, Wilcoxon rank-sum test; Hodges-Lehmann estimate = -0.25, 95% CI 2-sided [-0.50 to 0.00]
Statistical Analysis 3: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg BID (Period 1, 2 and 3); Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Hodges-Lehmann estimate = -0.50, 95% CI 2-sided [-0.75 to -0.25]

18. Secondary Outcome: Total Number of New or Enlarging T2 Lesions
Description: Analysis of New or Enlarging T2 lesions was done using magnetic resonance imaging (MRI) scans. As per planned analysis, Tecfidera treatment group was not included in inferential analysis.
Time Frame: Week 12 to Week 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 53 | 50 | 51 | 53 | 54
Lesions | 5.96 (6.994) | 6.52 (11.569) | 3.41 (10.752) | 2.19 (4.719) | 5.35 (16.667)
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Evobrutinib 25 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.4807, Negative Binomial; Lesion Rate ratio = 1.29, 95% CI 2-sided [0.63 to 2.65]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.0620, Negative Binomial; Lesion Rate ratio = 0.50, 95% CI 2-sided [0.24 to 1.04]
Statistical Analysis 3: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg BID (Period 1, 2 and 3); Test type: Superiority; p = 0.0189, Negative Binomial; Lesion Rate ratio = 0.42, 95% CI 2-sided [0.20 to 0.87]

19. Secondary Outcome: Change From Baseline in Volume of T2 Lesions at Week 24
Description: Analysis of volume of T2 lesions was done using magnetic resonance imaging (MRI) scans. Tecfidera treatment group was not included in inferential analysis.
Time Frame: Baseline, Week 24
Population: mITT analysis set consists of all participants who belong to both the ITT and safety analysis sets, and who have at least one baseline and one post-baseline magnetic resonance imaging (MRI) assessment. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cubic centimeter (cc)
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 44 | 46 | 48 | 46 | 50
cubic centimeter (cc) | 0.42 (1.009) | 0.93 (1.853) | -0.01 (0.562) | 0.09 (0.463) | 0.47 (2.964)
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Evobrutinib 25 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.8776, Mixed Effect Model for Repeat Measures; Difference in least squares means = 0.02, 95% CI 2-sided [-0.24 to 0.28] — Difference in least squares means of change from baseline in cube root of volume measured in centimeter
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.0019, Mixed Effect Model for Repeat Measures; Difference in least squares means = -0.41, 95% CI 2-sided [-0.66 to -0.15] — Difference in least squares means of change from baseline in cube root of volume measured in centimeter
Statistical Analysis 3: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg BID (Period 1, 2 and 3); Test type: Superiority; p = 0.0063, Mixed Effect Model for Repeat Measures; Difference in least squares means = -0.36, 95% CI 2-sided [-0.62 to -0.10] — Difference in least squares means of change from baseline in cube root of volume measured in centimeter

20. Secondary Outcome: Change From Baseline in Volume of Gadolinium-positive (Gd+) T1 Lesions at Week 24
Description: Analysis of volume of Gd+ T1 lesions was done using magnetic resonance imaging (MRI) scans. As per planned analysis, Tecfidera treatment group was not included in inferential analysis.
Time Frame: Baseline, Week 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Placebo (Period 1) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 53 | 50 | 51 | 53 | 54
cc | -0.023 (0.2220) | 0.057 (0.3479) | -0.111 (0.5416) | -0.051 (0.1032) | -0.050 (0.4771)
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Evobrutinib 25 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.9315, Wilcoxon rank-sum test; Hodges-Lehmann estimate = 0.00, 95% CI 2-sided [-0.004 to 0.009]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg QD (Period 1, 2 and 3); Test type: Superiority; p = 0.0008, Wilcoxon rank-sum test; Hodges-Lehmann estimate = -0.014, 95% CI 2-sided [-0.050 to 0.000]
Statistical Analysis 3: Comparison: Placebo (Period 1) vs Evobrutinib 75 mg BID (Period 1, 2 and 3); Test type: Superiority; p = 0.0014, Wilcoxon rank-sum test; Hodges-Lehmann estimate = -0.018, 95% CI 2-sided [-0.042 to 0.000]

21. Secondary Outcome: Number of Gadolinium-positive (Gd+) T1 Lesions at Week 48
Description: Analysis of Gd+ T1 lesions was done using magnetic resonance imaging (MRI) scans.
Time Frame: Week 48
Population: mITT BE analysis set included all participants who belonged to the mITT analysis set with an MRI assessment during the 24-week blinded extension period.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 44 | 44 | 46 | 45 | 50
Lesions | 1.00 (1.614) | 1.91 (4.296) | 0.85 (2.867) | 0.49 (1.218) | 0.42 (1.444)

22. Secondary Outcome: Number of New Gadolinium-positive (Gd+) T1 Lesions at Week 48
Description: Analysis of new Gd+ T1 lesions was done using magnetic resonance imaging (MRI) scans.
Time Frame: Week 48
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 44 | 44 | 46 | 45 | 50
Lesions | 0.95 (1.569) | 1.84 (4.154) | 0.85 (2.867) | 0.49 (1.218) | 0.42 (1.444)

23. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: A qualifying relapse is defined as new, worsening or recurrent neurological symptoms attributed to Multiple Sclerosis (MS) that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days.
Time Frame: Week 0 to Week 48
Population: as for outcome 17
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 53 | 50 | 51 | 53 | 54
relapses per year | 0.37 [0.21 to 0.59] | 0.52 [0.33 to 0.78] | 0.25 [0.12 to 0.44] | 0.11 [0.04 to 0.25] | 0.14 [0.06 to 0.29]

24. Secondary Outcome: Qualified Relapse-free Status
Description: A qualifying relapse is defined as new, worsening or recurrent neurological symptoms attributed to Multiple Sclerosis (MS) that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. Percentage of participants with qualified relapse-free status were reported.
Time Frame: Week 25 to Week 48
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 44 | 44 | 46 | 45 | 50
percentage of participants | 84.1 | 86.4 | 78.3 | 91.1 | 96.0

25. Secondary Outcome: Change From Week 24 in Expanded Disability Status Scale (EDSS) at Week 48
Description: The EDSS is an ordinal clinical rating scale in half-point increments. It assesses the following eight functional systems, areas of the central nervous system that control bodily functions: Pyramidal (ability to walk), Cerebellar (coordination), Brain stem (speech and swallowing), Sensory (touch and pain), Bowel and bladder functions, Visual, Mental, Other (includes any other neurological findings due to Multiple Sclerosis [MS]). EDSS overall score ranging from 0 (normal) to 10 (death due to MS).
Time Frame: Week 24, Week 48
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 44 | 44 | 46 | 45 | 50
Units on a scale | -0.05 (0.260) | -0.10 (0.351) | -0.01 (0.619) | 0.00 (0.238) | -0.10 (0.404)

26. Secondary Outcome: Total Number of New or Enlarging T2 Lesions at Week 48 Relative to Week 24
Description: Analysis of New or Enlarging T2 lesions was done using magnetic resonance imaging (MRI) scans.
Time Frame: Week 24 to Week 48
Population: mITT BE analysis set included all participants who belonged to the mITT analysis set with an MRI assessment during the 24-week blinded extension period. Here, "Number of Participants Analyzed" signified those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 42 | 42 | 43 | 43 | 50
Lesions | 3.57 (4.346) | 5.86 (11.330) | 3.84 (10.083) | 1.60 (3.799) | 1.88 (4.796)

27. Secondary Outcome: Change From Week 24 in Volume of Gadolinium-positive (Gd+) T1 Lesions at Week 48
Description: Analysis of volume of Gd+ T1 lesions was done using magnetic resonance imaging (MRI) scans.
Time Frame: Week 24, Week 48
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 44 | 44 | 46 | 45 | 50
cc | 0.092 (0.4626) | 0.088 (0.4006) | 0.045 (0.2285) | 0.024 (0.1981) | -0.203 (1.1073)

28. Secondary Outcome: Change From Week 24 in Volume of T2 Lesions at Week 48
Description: Analysis of volume of T2 lesions was done using magnetic resonance imaging (MRI) scans.
Time Frame: Week 24, Week 48
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 44 | 44 | 46 | 45 | 50
cc | 0.53 (1.360) | 0.67 (1.865) | 0.35 (1.083) | -0.03 (1.031) | -0.57 (2.699)

29. Secondary Outcome: OLE Period: Total Number of Gadolinium-Enhancing T1 Lesions
Description: Analysis of T1-Gadolinium enhancing lesions was done using magnetic resonance imaging (MRI) scans.
Time Frame: OLE Baseline (BE period Week 48), OLE Weeks 96, 144, 192, 240, 288 and 336
Population: modified ITT OLE Analysis Set (mITT-OLE) Analysis Set: participants randomly allocated to a treatment who belong to Safety OLE Analysis Set, and who have at least 1 Magnetic Resonance Imaging (MRI) assessment on or after OLE Week 0. Overall Number of Participants Analyzed= Participants evaluable for this outcome measure and Number analyzed= participants who were evaluable for the specified category. Results reported are for OLE period only and no participants took placebo during this period.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 34 | 35 | 37 | 44 | 37
Lesions
  OLE Baseline (BE period Week 48) | 0.82 (2.668) | 1.74 (4.395) | 1.46 (4.519) | 1.16 (3.050) | 2.03 (11.829)
  Week 96: number analyzed (Participants) | 31 | 27 | 35 | 36 | 36
  Week 96 | 0.13 (0.341) | 0.63 (1.822) | 0.49 (1.121) | 0.69 (1.411) | 0.67 (2.255)
  Week 144: number analyzed (Participants) | 29 | 27 | 34 | 35 | 31
  Week 144 | 0.76 (2.294) | 0.41 (1.217) | 0.82 (3.512) | 0.54 (1.146) | 1.29 (5.940)
  Week 192: number analyzed (Participants) | 28 | 25 | 32 | 32 | 26
  Week 192 | 1.00 (3.367) | 0.64 (1.890) | 0.81 (2.206) | 0.84 (1.798) | 0.96 (3.130)
  Week 240: number analyzed (Participants) | 25 | 24 | 30 | 30 | 26
  Week 240 | 1.68 (5.800) | 0.63 (1.996) | 0.37 (1.189) | 0.77 (2.417) | 0.88 (3.204)
  Week 288: number analyzed (Participants) | 20 | 17 | 28 | 26 | 23
  Week 288 | 0.35 (0.671) | 0.35 (0.786) | 0.32 (1.090) | 1.04 (2.946) | 0.35 (1.265)
  Week 336: number analyzed (Participants) | 6 | 7 | 6 | 7 | 15
  Week 336 | 0.83 (1.602) | 3.00 (5.745) | 1.17 (2.858) | 0.29 (0.756) | 5.60 (18.310)

30. Secondary Outcome: OLE Period: Annualized Relapse Rate (ARR)
Description: as for outcome 23
Time Frame: OLE Baseline (BE period Week 48), OLE Weeks 96, 144, 192, 240, 288 and 336
Population: modified ITT OLE Analysis Set (mITT-OLE) Analysis Set: participants randomly allocated to a treatment who belong to Safety OLE Analysis Set, and who have at least 1 Magnetic Resonance Imaging (MRI) assessment on or after OLE Week 0. Here, "Number analyzed" signifies those participants who were evaluable for the specified category. Results reported are for OLE period only and no participants took placebo during this period.
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 39 | 38 | 42 | 44 | 48
relapses per year
  OLE Baseline (BE period Week 48) | 0.29 [0.14 to 0.53] | 0.18 [0.06 to 0.38] | 0.14 [0.04 to 0.32] | 0.17 [0.07 to 0.36] | 0.12 [0.04 to 0.28]
  Week 96: number analyzed (Participants) | 37 | 36 | 37 | 44 | 40
  Week 96 | 0.16 [0.05 to 0.37] | 0.13 [0.04 to 0.34] | 0.09 [0.02 to 0.26] | 0.08 [0.02 to 0.22] | 0.03 [0.00 to 0.16]
  Week 144: number analyzed (Participants) | 33 | 30 | 37 | 40 | 36
  Week 144 | 0.07 [0.01 to 0.25] | 0.11 [0.02 to 0.33] | 0.03 [0.00 to 0.17] | 0.15 [0.05 to 0.34] | 0.16 [0.05 to 0.37]
  Week 192: number analyzed (Participants) | 31 | 27 | 35 | 35 | 33
  Week 192 | 0.04 [0.00 to 0.20] | 0.08 [0.01 to 0.29] | 0.22 [0.09 to 0.45] | 0.16 [0.05 to 0.38] | 0.04 [0.00 to 0.20]
  Week 240: number analyzed (Participants) | 30 | 27 | 34 | 33 | 30
  Week 240 | 0.16 [0.04 to 0.41] | 0.04 [0.00 to 0.23] | 0.10 [0.02 to 0.28] | 0.13 [0.04 to 0.34] | 0.00 [NA to 0.15] — Based on pre-specified criteria, when the number of qualified relapses is zero, the lower limit of 95% confidence interval could not be calculated.
  Week 288: number analyzed (Participants) | 25 | 24 | 32 | 32 | 26
  Week 288 | 0.13 [0.13 to 0.38] | 0.05 [0.00 to 0.25] | 0.07 [0.01 to 0.25] | 0.00 [NA to 0.13] — Based on pre-specified criteria, when the number of qualified relapses is zero, the lower limit of 95% confidence interval could not be calculated. | 0.04 [0.00 to 0.24]
  Week 336: number analyzed (Participants) | 24 | 22 | 26 | 29 | 7
  Week 336 | 0.00 [NA to 1.75] — Based on pre-specified criteria, when the number of qualified relapses is zero, the lower limit of 95% confidence interval could not be calculated. | 0.00 [NA to 1.55] — Based on pre-specified criteria, when the number of qualified relapses is zero, the lower limit of 95% confidence interval could not be calculated. | 0.31 [0.01 to 1.70] | 0.00 [NA to 1.27] — Based on pre-specified criteria, when the number of qualified relapses is zero, the lower limit of 95% confidence interval could not be calculated. | 0.00 [NA to 7.97] — Based on pre-specified criteria, when the number of qualified relapses is zero, the lower limit of 95% confidence interval could not be calculated.

31. Secondary Outcome: OLE Period: Percentage of Participants With Qualified Relapse-Free Status
Description: A qualifying relapse is defined as new, worsening or recurrent neurological symptoms attributed to Multiple Sclerosis (MS) that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. Percentage of participants with qualified relapse-free status from OLE Baseline (BE period Week 48) up to Week 336 were reported.
Time Frame: OLE Baseline (BE period Week 48) up to OLE Week 336
Population: modified ITT OLE Analysis Set (mITT-OLE) Analysis Set: participants randomly allocated to a treatment who belong to Safety OLE Analysis Set, and who have at least 1 Magnetic Resonance Imaging (MRI) assessment on or after OLE Week 0. Overall Number of Participants Analyzed= Participants evaluable for this outcome measure. Results reported are for OLE period only and no participants took placebo during this period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 39 | 38 | 42 | 44 | 48
percentage of participants | 66.7 | 68.4 | 71.4 | 65.9 | 83.3

32. Secondary Outcome: OLE Period: Change From Baseline in Expanded Disability Status Scale (EDSS) at Week 96, 144, 192, 240, 288 and 336
Description: as for outcome 25
Time Frame: OLE Baseline (BE period Week 48), OLE Weeks 96, 144, 192, 240, 288 and 336
Population: modified ITT OLE Analysis Set (mITT-OLE) Analysis Set: participants randomly allocated to a treatment who belong to Safety OLE Analysis Set, and who have at least 1 Magnetic Resonance Imaging (MRI) assessment on or after OLE Week 0. Overall Number of Participants Analyzed= Participants evaluable for this outcome measure and Number analyzed = participants who were evaluable for the specified category. Results reported are for OLE period only and no participants took placebo during this period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 39 | 38 | 42 | 44 | 48
units on a scale
  OLE Baseline (BE period Week 48): number analyzed (Participants) | 37 | 35 | 28 | 44 | 40
  OLE Baseline (BE period Week 48) | 0.1 (0.39) | 0.0 (0.69) | 0.1 (0.46) | 0.0 (0.27) | 0.0 (0.34)
  Week 96: number analyzed (Participants) | 34 | 30 | 35 | 38 | 36
  Week 96 | 0.1 (0.40) | 0.1 (0.46) | 0.2 (0.71) | 0.0 (0.42) | 0.0 (0.32)
  Week 144: number analyzed (Participants) | 31 | 27 | 36 | 35 | 32
  Week 144 | 0.1 (0.79) | 0.1 (0.61) | 0.2 (0.79) | 0.0 (0.44) | 0.0 (0.28)
  Week 192: number analyzed (Participants) | 28 | 26 | 34 | 33 | 28
  Week 192 | 0.2 (0.64) | 0.1 (0.61) | 0.2 (0.35) | 0.2 (0.72) | 0.0 (0.29)
  Week 240: number analyzed (Participants) | 25 | 25 | 32 | 32 | 26
  Week 240 | 0.3 (0.72) | 0.3 (0.50) | 0.2 (0.46) | 0.2 (0.93) | 0.1 (0.40)
  Week 288: number analyzed (Participants) | 23 | 23 | 29 | 29 | 25
  Week 288 | 0.4 (0.80) | 0.1 (0.87) | 0.4 (0.58) | 0.4 (0.81) | 0.2 (0.45)
  Week 336: number analyzed (Participants) | 11 | 10 | 10 | 7 | 15
  Week 336 | 0.0 (0.52) | 0.5 (1.36) | 0.7 (1.38) | -0.2 (0.57) | 0.0 (0.52)

33. Secondary Outcome: OLE Period: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: as for outcome 5
Time Frame: OLE Baseline (BE period Week 48) up to OLE Week 336
Population: The Safety OLE Analysis Set included all participants who receive at least 1 dose of Evobrutinib during the OLE. Results reported are for OLE period only and no participants took placebo during this period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 39 | 39 | 42 | 44 | 49
Participants | 35 | 29 | 41 | 40 | 37

34. Secondary Outcome: OLE Period: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Vital signs, including semi supine blood pressure, pulse rate, respiratory rate, weight, and oral temperature were assessed. Number of participants with clinically significant change from baseline in vital signs were reported. Clinical Significance was decided by the investigator.
Time Frame: OLE Baseline (BE period Week 48) up to OLE Week 336
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 39 | 39 | 42 | 44 | 49
Participants | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: OLE Period: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameters
Description: Laboratory parameters included hematology, biochemistry, and urinalysis. Number of participants with clinically significant change from baseline in laboratory parameters were reported. Clinical Significance was decided by the investigator.
Time Frame: OLE Baseline (BE period Week 48) up to OLE Week 336
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 39 | 39 | 42 | 44 | 49
Participants | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: OLE Period: Number of Participants With Clinically Significant Changes From Baseline in Electrocardiograms (ECGs)
Description: ECG parameters included rhythm, ventricular rate, PR interval, QRS duration, and QT interval. Number of participants with clinically significant change from baseline in ECG were reported. Clinical Significance was decided by the investigator.
Time Frame: OLE Baseline (BE period Week 48) up to OLE Week 336
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 39 | 39 | 42 | 44 | 49
Participants | 0 | 0 | 0 | 0 | 0

37. Secondary Outcome: OLE Period: Absolute Concentrations of Immunoglobulin (Ig) Levels
Description: Absolute Concentrations serum levels of IgG, IgA, IgM were assessed.
Time Frame: OLE Baseline (BE period Week 48), OLE Weeks 96, 144, 192, 240 and 288
Population: The Safety OLE Analysis Set included all participants who receive at least 1 dose of Evobrutinib during the OLE. Overall Number of Participants Analyzed= Participants evaluable for this outcome measure and Number analyzed = participants who were evaluable for the specified category. Results reported are for OLE period only and no participants took placebo during this period.
Measure: Mean (Standard Deviation); unit: Gram per Liter
Arm/Group | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 37 | 37 | 37 | 44 | 40
Gram per Liter
  Ig A, OLE Baseline (BE period Week 48) | 2.31 (0.966) | 2.44 (0.897) | 2.49 (0.953) | 2.52 (0.970) | 2.31 (0.906)
  Ig A, Week 72: number analyzed (Participants) | 34 | 32 | 35 | 43 | 37
  Ig A, Week 72 | 2.38 (1.084) | 2.53 (1.075) | 2.72 (1.137) | 2.65 (1.062) | 2.43 (0.865)
  Ig A, Week 96: number analyzed (Participants) | 32 | 30 | 36 | 39 | 38
  Ig A, Week 96 | 2.42 (1.173) | 2.69 (1.026) | 2.91 (1.181) | 2.82 (1.113) | 2.62 (1.072)
  Ig A, Week 144: number analyzed (Participants) | 30 | 27 | 36 | 35 | 33
  Ig A, Week 144 | 2.57 (1.274) | 2.73 (0.918) | 2.82 (1.326) | 2.91 (1.233) | 2.57 (1.025)
  IgA, Week 192: number analyzed (Participants) | 29 | 26 | 33 | 32 | 26
  IgA, Week 192 | 2.60 (1.242) | 2.71 (0.987) | 2.86 (1.255) | 3.15 (1.185) | 2.70 (1.055)
  IgA, Week 240: number analyzed (Participants) | 24 | 22 | 33 | 28 | 23
  IgA, Week 240 | 2.71 (1.280) | 2.85 (1.095) | 3.05 (1.314) | 3.13 (1.269) | 2.65 (0.984)
  IgA, Week 288: number analyzed (Participants) | 37 | 20 | 26 | 27 | 17
  IgA, Week 288 | 2.68 (1.305) | 3.08 (1.276) | 3.12 (1.306) | 3.30 (1.347) | 2.92 (1.108)
  Ig G, OLE Baseline (BE period Week 48) | 9.75 (2.253) | 10.37 (2.512) | 10.73 (2.479) | 10.44 (2.291) | 9.65 (2.165)
  Ig G, Week 72: number analyzed (Participants) | 34 | 32 | 35 | 43 | 37
  Ig G, Week 72 | 9.63 (2.335) | 10.47 (2.509) | 10.69 (2.515) | 10.42 (2.116) | 9.93 (2.131)
  Ig G, Week 96: number analyzed (Participants) | 32 | 30 | 36 | 39 | 38
  Ig G, Week 96 | 9.46 (2.490) | 10.10 (2.461) | 10.76 (2.413) | 10.29 (2.172) | 9.93 (2.285)
  Ig G, Week 144: number analyzed (Participants) | 30 | 27 | 36 | 35 | 33
  Ig G, Week 144 | 9.48 (2.294) | 10.43 (2.304) | 10.38 (2.638) | 10.21 (2.552) | 9.32 (2.115)
  IgG, Week 192: number analyzed (Participants) | 29 | 26 | 33 | 32 | 26
  IgG, Week 192 | 9.37 (2.156) | 9.99 (2.197) | 10.36 (2.548) | 10.46 (2.135) | 9.56 (2.094)
  IgG, Week 240: number analyzed (Participants) | 24 | 22 | 33 | 28 | 23
  IgG, Week 240 | 9.28 (2.081) | 10.33 (2.422) | 10.47 (2.562) | 10.47 (2.562) | 9.58 (2.245)
  IgG, Week 288: number analyzed (Participants) | 25 | 20 | 26 | 27 | 17
  IgG, Week 288 | 9.46 (2.068) | 10.48 (2.541) | 10.64 (2.566) | 10.36 (2.273) | 9.72 (2.700)
  Ig M, OLE Baseline (BE period Week 48) | 1.06 (0.550) | 0.89 (0.403) | 1.08 (0.680) | 0.92 (0.422) | 0.99 (0.586)
  Ig M, Week 72: number analyzed (Participants) | 34 | 32 | 35 | 43 | 37
  Ig M, Week 72 | 1.03 (0.551) | 0.87 (0.397) | 1.05 (0.758) | 0.91 (0.425) | 0.94 (0.561)
  Ig M, Week 96: number analyzed (Participants) | 32 | 30 | 36 | 39 | 38
  Ig M, Week 96 | 1.01 (0.556) | 0.87 (0.413) | 1.05 (0.747) | 0.92 (0.460) | 0.91 (0.525)
  Ig M, Week 144: number analyzed (Participants) | 30 | 27 | 36 | 35 | 33
  Ig M, Week 144 | 0.88 (0.463) | 0.88 (0.468) | 0.94 (0.614) | 0.89 (0.377) | 0.90 (0.519)
  Ig M, Week 192: number analyzed (Participants) | 28 | 26 | 33 | 32 | 26
  Ig M, Week 192 | 0.89 (0.492) | 0.87 (0.461) | 0.90 (0.462) | 0.84 (0.320) | 0.90 (0.585)
  Ig M, Week 240: number analyzed (Participants) | 24 | 22 | 33 | 28 | 23
  Ig M, Week 240 | 0.85 (0.420) | 0.83 (0.419) | 0.87 (0.468) | 0.88 (0.369) | 0.87 (0.611)
  Ig M, Week 288: number analyzed (Participants) | 25 | 22 | 27 | 28 | 18
  Ig M, Week 288 | 0.85 (0.405) | 0.90 (0.490) | 0.94 (0.544) | 0.87 (0.397) | 1.03 (0.568)

38. Secondary Outcome: OLE Period: Change From Baseline in Immunoglobulin (Ig) Levels
Description: Change from baseline in the serum levels of IgG, IgA, IgM were assessed.
Time Frame: OLE Baseline (BE period Week 48), OLE Weeks 96, 144, 192, 240 and 288
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Gram per Liter
Arm/Group | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg QD (Period 1, 2 and 3) | Evobrutinib 75 mg BID (Period 1, 2 and 3) | Tecfidera (Period 1, 2 and 3)
Number analyzed (Participants) | 37 | 37 | 37 | 44 | 40
Gram per Liter
  Ig A, OLE Baseline (BE period Week 48) | 0.26 (0.237) | 0.17 (0.333) | 0.19 (0.283) | 0.26 (0.291) | 0.28 (0.355)
  Ig A, Week 72: number analyzed (Participants) | 34 | 32 | 35 | 43 | 37
  Ig A, Week 72 | 0.40 (0.398) | 0.36 (0.515) | 0.41 (0.417) | 0.38 (0.453) | 0.42 (0.368)
  Ig A, Week 96: number analyzed (Participants) | 32 | 30 | 36 | 39 | 38
  Ig A, Week 96 | 0.44 (0.491) | 0.45 (0.407) | 0.58 (0.485) | 0.54 (0.446) | 0.59 (0.545)
  Ig A, Week 144: number analyzed (Participants) | 30 | 27 | 36 | 35 | 33
  Ig A, Week 144 | 0.58 (0.594) | 0.41 (0.347) | 0.50 (0.670) | 0.57 (0.589) | 0.54 (0.452)
  IgA, Week 192: number analyzed (Participants) | 29 | 26 | 33 | 32 | 26
  IgA, Week 192 | 0.60 (0.597) | 0.38 (0.443) | 0.55 (0.667) | 0.82 (0.530) | 0.67 (0.492)
  IgA, Week 240: number analyzed (Participants) | 24 | 22 | 33 | 28 | 23
  IgA, Week 240 | 0.67 (0.605) | 0.55 (0.471) | 0.74 (0.682) | 0.78 (0.621) | 0.68 (0.520)
  IgA, Week 288: number analyzed (Participants) | 25 | 20 | 26 | 27 | 17
  IgA, Week 288 | 0.68 (0.934) | 0.75 (0.680) | 0.91 (0.915) | 1.02 (0.637) | 0.93 (0.724)
  Ig G, OLE Baseline (BE period Week 48) | 0.39 (0.960) | 0.54 (1.463) | 0.69 (1.147) | 1.11 (1.150) | 0.23 (1.216)
  Ig G, Week 72: number analyzed (Participants) | 34 | 32 | 35 | 43 | 37
  Ig G, Week 72 | 0.40 (1.019) | 0.56 (1.364) | 0.79 (1.236) | 1.07 (0.994) | 0.48 (1.288)
  Ig G, Week 96: number analyzed (Participants) | 32 | 30 | 36 | 39 | 38
  Ig G, Week 96 | 0.17 (1.359) | 0.18 (1.228) | 0.64 (1.178) | 0.84 (1.073) | 0.47 (1.355)
  Ig G, Week 144: number analyzed (Participants) | 30 | 27 | 36 | 35 | 33
  Ig G, Week 144 | 0.35 (1.367) | 0.17 (1.451) | 0.31 (1.356) | 0.68 (1.458) | -0.09 (1.176)
  IgG, Week 192: number analyzed (Participants) | 29 | 26 | 33 | 32 | 26
  IgG, Week 192 | 0.14 (1.227) | -0.13 (1.141) | 0.18 (1.625) | 0.84 (1.384) | 0.09 (1.324)
  IgG, Week 240: number analyzed (Participants) | 24 | 22 | 33 | 28 | 23
  IgG, Week 240 | -0.01 (1.336) | 0.10 (1.557) | 0.37 (1.596) | 0.75 (1.362) | 0.19 (1.314)
  IgG, Week 288: number analyzed (Participants) | 25 | 20 | 26 | 27 | 17
  IgG, Week 288 | 0.18 (1.492) | 0.48 (1.465) | 0.37 (2.203) | 1.01 (1.570) | 0.36 (1.440)
  Ig M, OLE Baseline (BE period Week 48) | -0.18 (0.152) | -0.10 (0.120) | -0.09 (0.122) | -0.05 (0.099) | -0.28 (0.280)
  IgM, Week 72: number analyzed (Participants) | 34 | 32 | 35 | 43 | 37
  IgM, Week 72 | -0.19 (0.170) | -0.11 (0.119) | -0.10 (0.147) | -0.07 (0.104) | -0.34 (0.264)
  IgM, Week 96: number analyzed (Participants) | 32 | 30 | 36 | 39 | 38
  IgM, Week 96 | -0.23 (0.146) | -0.13 (0.141) | -0.09 (0.199) | -0.08 (0.127) | -0.35 (0.301)
  IgM, Week 144: number analyzed (Participants) | 30 | 27 | 36 | 35 | 33
  IgM, Week 144 | -0.28 (0.323) | -0.14 (0.195) | -0.17 (0.174) | -0.11 (0.149) | -0.40 (0.327)
  IgM, Week 192: number analyzed (Participants) | 28 | 26 | 33 | 32 | 26
  IgM, Week 192 | -0.28 (0.254) | -0.16 (0.204) | -0.19 (0.186) | -0.18 (0.197) | -0.46 (0.330)
  IgM, Week 240: number analyzed (Participants) | 24 | 22 | 33 | 28 | 23
  IgM, Week 240 | -0.29 (0.282) | -0.20 (0.187) | -0.19 (0.205) | -0.16 (0.254) | -0.53 (0.348)
  IgM, Week 288: number analyzed (Participants) | 25 | 22 | 27 | 28 | 18
  IgM, Week 288 | -0.29 (0.284) | -0.11 (0.313) | -0.15 (0.315) | -0.17 (0.178) | -0.39 (0.472)

ADVERSE EVENTS:
Time Frame: Baseline up to Safety Follow up of blinded extension period (Week 52); OLE Baseline (BE period Week 48) up to OLE Week 336
Description: Active treatment period and BE period: MedDRA version 21.0; OLE Period: MedDRA version 26.1
Groups:
- Evobrutinib 25 mg QD (Period 1 and Period 2): Participants received Evobrutinib 25 mg orally, QD up to Week 48 in active treatment period 1 and BE period.
- Evobrutinib 75 mg QD (Period 1 and Period 2): Participants received Evobrutinib 75 mg orally, QD up to Week 48 in active treatment period 1 and BE period.
- Evobrutinib 75 mg BID (Period 1 and Period 2): Participants received Evobrutinib 75 mg orally, twice daily (BID) up to Week 48 in active treatment period 1 and BE period.
- Tecfidera (Period 1 and Period 2): Participants received Tecfidera 120 mg twice daily (BID) for first 7 days followed by 240 mg orally, BID up to Week 48 in active treatment period 1 and BE period.
- Evobrutinib 25 mg QD (Period 3): Participants received Evobrutinib 25 mg QD orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
- Evobrutinib 75 mg QD (Period 3): Participants received Evobrutinib 75 mg QD orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
- Evobrutinib 75 mg BID (Period 3): Participants received Evobrutinib 75 mg BID orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
- Tecfidera (Period 3): Participants received Tecfidera 120 mg BID orally from Week 48 of BE period (OLE period Day 1) to Week 336 in OLE period.
Arm/Group | Placebo (Period 1) | Placebo Then Evobrutinib 25 mg QD (Period 2) | Evobrutinib 25 mg QD (Period 1 and Period 2) | Evobrutinib 75 mg QD (Period 1 and Period 2) | Evobrutinib 75 mg BID (Period 1 and Period 2) | Tecfidera (Period 1 and Period 2) | Placebo + Evobrutinib 25 mg QD (Period 3) | Evobrutinib 25 mg QD (Period 3) | Evobrutinib 75 mg QD (Period 3) | Evobrutinib 75 mg BID (Period 3) | Tecfidera (Period 3)
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/49 | 0/52 | 0/53 | 0/54 | 0/54 | 0/39 | 1/39 | 0/42 | 1/44 | 1/49
Serious Adverse Events (participants affected / at risk) | 2/54 | 0/49 | 2/52 | 2/53 | 4/54 | 2/54 | 7/39 | 12/39 | 8/42 | 5/44 | 10/49
Other Adverse Events (participants affected / at risk) | 14/54 | 9/49 | 19/52 | 19/53 | 20/54 | 30/54 | 30/39 | 26/39 | 34/42 | 31/44 | 26/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Period 1) (N=54) | Placebo Then Evobrutinib 25 mg QD (Period 2) (N=49) | Evobrutinib 25 mg QD (Period 1 and Period 2) (N=52) | Evobrutinib 75 mg QD (Period 1 and Period 2) (N=53) | Evobrutinib 75 mg BID (Period 1 and Period 2) (N=54) | Tecfidera (Period 1 and Period 2) (N=54) | Placebo + Evobrutinib 25 mg QD (Period 3) (N=39) | Evobrutinib 25 mg QD (Period 3) (N=39) | Evobrutinib 75 mg QD (Period 3) (N=42) | Evobrutinib 75 mg BID (Period 3) (N=44) | Tecfidera (Period 3) (N=49)
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keratoconus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Serratia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebellar ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Multiple sclerosis pseudo relapse (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertebrobasilar artery dissection (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo CNS origin (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bladder hypertrophy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uterine cervix stenosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Period 1) (N=54) | Placebo Then Evobrutinib 25 mg QD (Period 2) (N=49) | Evobrutinib 25 mg QD (Period 1 and Period 2) (N=52) | Evobrutinib 75 mg QD (Period 1 and Period 2) (N=53) | Evobrutinib 75 mg BID (Period 1 and Period 2) (N=54) | Tecfidera (Period 1 and Period 2) (N=54) | Placebo + Evobrutinib 25 mg QD (Period 3) (N=39) | Evobrutinib 25 mg QD (Period 3) (N=39) | Evobrutinib 75 mg QD (Period 3) (N=42) | Evobrutinib 75 mg BID (Period 3) (N=44) | Tecfidera (Period 3) (N=49)
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 3 | 3 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 3
Nasopharyngitis (Infections and infestations) | 5 | 1 | 9 | 3 | 7 | 2 | 7 | 7 | 8 | 9 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 3 | 5 | 2 | 6 | 4 | 3
Alanine aminotransferase increased (Investigations) | 3 | 1 | 3 | 6 | 5 | 3 | 1 | 1 | 0 | 0 | 5
Lipase increased (Investigations) | 2 | 3 | 2 | 5 | 5 | 3 | 5 | 6 | 6 | 8 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 3 | 3 | 1 | 2 | 1 | 2 | 3 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1 | 3 | 1 | 2 | 0 | 1 | 0 | 3
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 2 | 0 | 1 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3 | 0 | 4 | 5 | 3 | 1 | 2 | 2
Headache (Nervous system disorders) | 2 | 0 | 3 | 2 | 1 | 1 | 3 | 2 | 5 | 6 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 2 | 1 | 0 | 0 | 7 | 5 | 7 | 5 | 3
Cystitis (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 1 | 0
Vaccination site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 3 | 6 | 7
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 1 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 9 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 3 | 1 | 3
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 2

LIMITATIONS AND CAVEATS:
Reported p values are not adjusted for multiple testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT02975349/Prot_002.pdf
  • Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT02975349/SAP_003.pdf